CLINICAL TRIAL: NCT01749475
Title: Hypnosis for Sedation in Transesophageal Echocardiography: Comparison With Midazolam
Brief Title: Hypnosis vs Midazolam for Sedation for TEE
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYPTEE
Record Dates: First submitted 2012-12-12; First posted 2012-12-13 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Clinical Indications for Transesophageal Echocardiography
MeSH Terms: interventions — Midazolam; Hypnosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- midazolam
  Interventions: Drug: Midazolam
- hypnosis
  Interventions: Other: hypnotherapy

INTERVENTIONS:
Drug: Midazolam — The patients will be given 0.05mg/kg iv midazolam just before monitorization. During probing, in case of intolerance to the insertion of the probe, the increments of midazolam with 0.005mg/kg doses will be given.
  Groups: midazolam
Other: hypnotherapy — A first hypnotic induction will be carried out the day before the procedure, next day, fifteen minutes before the procedure, a new induction will be performed.
  Groups: hypnosis

SUMMARY:
Most of the reports on hypnosis in the literature have focused on pain control during minor operations. With this study we aimed to evaluate the role of hypnosis on sedation for transesophageal echocardiography and compare it with commonly used sedative midazolam.

ELIGIBILITY:
Inclusion Criteria:

* indications for TEE
* American Society of Anesthesiology (ASA) physical status I-III

Exclusion Criteria:

* mental illness,
* psychotropic medication use,
* hypersensitivity to drugs
* a body mass index over 30.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitting to cardiology department for transesophageal echocardiography (TEE)
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-06; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Sedative effects of hypnotherapy and the drug "midazolam" indicated by anxiety scores and bispectral index (BIS) monitoring | during transesophageal echocardiography

SECONDARY OUTCOMES:
measurement of alertness after sedation with continuous performance test (CPT) | the same time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi Konuk Training Hospital, Istanbul, Turkey (Türkiye)